CLINICAL TRIAL: NCT00805311
Title: Carotid Endarterectomy Versus Optimal Medical Treatment of Asymptomatic High Grade Carotid Artery Stenosis
Brief Title: Aggressive Medical Treatment Evaluation for Asymptomatic Carotid Artery Stenosis
Acronym: AMTEC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the clear advantage of carotid endarterectomy
Sponsor: Russian Cardiology Research and Production Center (Other)
Responsible Party: Principal Investigator, Igor Kolos, Senior Researcher, Russian Cardiology Research and Production Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT00805311
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Carotid Artery Stenosis; Atherosclerosis; Stroke
Keywords: Internal Carotid Artery Stenosis; Carotid Endarterectomy; Stroke; Cerebrovascular; Atherosclerosis
MeSH Terms: conditions — Carotid Stenosis; Atherosclerosis; Stroke | interventions — Endarterectomy, Carotid; Atorvastatin; Aspirin; Losartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CEA Group (Experimental): Patients will undergo carotid endarterectomy (CEA) and receive medical treatment including medical therapy with statins (at least 10 mg atorvastatin irrespective of the baseline cholesterol level), aspirin (100 mg daily) and antihypertensive therapy (at least 50 mg losartan and 5 mg amlodipine 75 mg daily irrespective of the baseline arterial pressure level). Further conservative medical treatment includes modification of cardiovascular risk factors according to current recommendations.
  Interventions: Procedure: Carotid Endarterectomy; Drug: atorvastatin, aspirin, losartan, amlodipine
- OMT Group (Active Comparator): Patients will receive conservative therapy - optimal medical treatment (OMT) including statins (at least 10 mg atorvastatin irrespective of the baseline cholesterol level), aspirin (100 mg daily) and antihypertensive therapy (at least 50 mg losartan and 5 mg amlodipine 75 mg daily irrespective of the baseline arterial pressure level). Further conservative medical treatment includes modification of cardiovascular risk factors according to current recommendations.
  Interventions: Drug: atorvastatin, aspirin, losartan, amlodipine

INTERVENTIONS:
Procedure: Carotid Endarterectomy — CEA involves a neck incision and physical removal of the plaque from the inside of the artery
  Arms: CEA Group
Drug: atorvastatin, aspirin, losartan, amlodipine — aspirin 100 mg/day, atorvastatin 10 mg/day, losartan 50 mg/day, amlodipine 5 mg/day

SUMMARY:
The aim of this study is to determine whether optimal medical treatment can postpone carotid endarterectomy.

DETAILED DESCRIPTION:
It is well known that risk of fatal and non-fatal stroke is increased in patients with significant carotid atherosclerosis. For asymptomatic patients, AHA guidelines recommend carotid endarterectomy (CEA) for stenosis 60% to 99%, if the risk of perioperative stroke or death is less than 3%.

Although clinical trial data support CEA in asymptomatic patients with carotid stenosis 60% to 79%, the AHA guidelines indicate that some physicians delay revascularization until there is greater than 80% stenosis in asymptomatic patients.

Our study is designed to determine whether optimal medical therapy alone reduces the risk of death and nonfatal stroke in patients with carotid artery stenosis as compared with CEA coupled with optimal medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral carotid artery stenosis that was considered to be severe (carotid artery diameter reduction 70%-79% on ultrasound)
* This stenosis had not caused any stroke, transient cerebral ischaemia, or other relevant neurological symptoms in the past 6 months
* Both doctor and patient were substantially uncertain whether to choose immediate CEA, or deferral of any CEA until a more definite need for it was thought to have arisen
* The patient had no known circumstance or condition likely to preclude long-term follow-up
* Neurologist's explicit consent to potentially perform CEA

Exclusion Criteria:

* Previous ipsilateral CEA
* Expectation of poor surgical risk (e.g., because of recent acute myocardial infarction)
* Some probable cardiac source of emboli (because the main stroke risk might then be from cardiac, not carotid, emboli)
* Inability to provide informed consent
* Underlying disease other than atherosclerosis (inflammatory or autoimmune disease)
* Life expectancy < 6 months
* Advanced dementia
* Advanced renal failure (serum creatinine > 2.5 mg/dL)
* Unstable severe cardiovascular comorbidities (e.g., unstable angina, heart failure)
* Restenosis after prior CAS or CEA
* Atrial fibrillation
* Allergy or contraindications to study medications (statins, ASA, losartan, amlodipine)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
composite of nonfatal stroke, nonfatal composite of nonfatal stroke, nonfatal myocardial infarction and death | 5 years

SECONDARY OUTCOMES:
composite of nonfatal stroke, nonfatal MI, carotid/coronary revascularization and death | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniy Chazov, MD, Study Chair — Russian Cardiology Research and Production Center
Locations (1):
- Russian Cardiology Research and Production Center, Moscow, Russia

REFERENCES:
- [Background] Kolos I, Troitskiy A, Balakhonova T, Shariya M, Skrypnik D, Tvorogova T, Deev A, Boytsov S; Aggressive Medical Treatment Evaluation for Asymptomatic Carotid Artery Stenosis (AMTEC) Study Group. Modern medical treatment with or without carotid endarterectomy for severe asymptomatic carotid atherosclerosis. J Vasc Surg. 2015 Oct;62(4):914-22. doi: 10.1016/j.jvs.2015.05.005. PMID 26410046
- [Result] Kolos I, Loukianov M, Dupik N, Boytsov S, Deev A. Optimal medical treatment versus carotid endarterectomy: the rationale and design of the Aggressive Medical Treatment Evaluation for Asymptomatic Carotid Artery Stenosis (AMTEC) study. Int J Stroke. 2015 Feb;10(2):269-74. doi: 10.1111/ijs.12019. Epub 2013 Mar 15. PMID 23490405